CLINICAL TRIAL: NCT05380778
Title: BIS Controlled Anesthesia Depth is Associated With Different Protein and Peptide Expression in the Cerebrospinal Fluid
Brief Title: Depth of Anesthesia and Proteomics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Thomas Frietsch, Associate Professor, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TF-KliMa-2005-2
Record Dates: First submitted 2022-05-13; First posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia Complication; Immune Suppression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shallow Anesthesia (Experimental): Experimental: Shallow Anesthesia Standard anesthesia with fentanyl, propofol for shoulder surgery together with an interscalene plexus block was performed. The anesthesiologist only was informed about the group allocation by the study director and tried to control best for maintenance on target anesthesia level BIS ≥ 55 (group 2, shallow anesthesia). Anesthesia depth as measured by BIS monitors (BIS Vista, Aspect) for every minute and the minutes above a BIS level of 45 were counted.
  Interventions: Drug: Shallow anesthesia
- Deep Anesthesia (Experimental): Experimental: Deep Anesthesia Standard anesthesia with fentanyl, propofol for shoulder surgery together with an interscalene plexus block was performed. The anesthesiologist only was informed about the group allocation by the study director and tried to control best for maintenance on target anesthesia level BIS < 45 (group 1, deep anesthesia). Anesthesia depth as measured by BIS monitors (BIS Vista, Aspect) for every minute and the minutes below a BIS level of 45 were counted.
  Interventions: Drug: Deep anesthesia

INTERVENTIONS:
Drug: Deep anesthesia — Drug: High dose propofol, fentanyl and sevoflurane Deep Anesthesia
  Other Names:
  BIS lower than or equal to 45
  Other Names: Profound anesthesia
  Arms: Deep Anesthesia
Drug: Shallow anesthesia — Drug: Low dose propofol, fentanyl and sevoflurane Shallow Anesthesia
  Other Names:
  BIS above 45
  Other Names: Light anesthesia
  Arms: Shallow Anesthesia

SUMMARY:
The primary aim of the study is to compare cellular activity of T-cells, NK-cells and monocytes after anesthesia. Phagocytosis and cellular lysis activity of neutrophils and monocytes are analyzed by flow cytometry. Secondly, we analyze anesthesia induced protein expresssion pattern in the blood. The proteome of monocytes is identified by 3D-gel-chromatography and mass spectrometry (MALDI-TOF).

DETAILED DESCRIPTION:
Patients undergoing shoulder surgery in the orthopedic center are screened and consented to the randomized controlled, blinded study. Patients, surgeons, and the study personell involved in data interpretation and management are blinded towards the randomly assigned computerized group allocation (SAS, Cary, NC). The study director informs the anesthesiology staff about the group allocation. Patients are randomized to deep vs. light general anesthesia guided using a bispectral index monitor (BIS Vista, Aspect) with BIS < 45 in group 1 (deep anesthesia) or BIS ≥ 55 in group 2 (light anesthesia). Anesthesia depth is recorded via USB port every minute.

ELIGIBILITY:
Inclusion Criteria:

enrolment for longer shoulder surgery consent for the standard anesthesia form in combination with the interscalene plexus block ASA Status 1-3

Exclusion Criteria:

sedative premedication severe immune deficiency (diabetes, steroid or antihistamine medication, cancer, chemotherapy, status post transplantation, drug and alcohol abuse), recent surgery (1 month) or blood transfusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-03-01 (Actual); Primary Completion 2014-07-15 (Actual); Study Completion 2016-10-23 (Actual)

PRIMARY OUTCOMES:
Proteome: depression of immune stimulative proteins | 70-90 min
  Primary Outcome Measure:
  1.Depression of immune stimulating proteins in the proteom of maccrophages in in the 3-D- Gel electrophoresis as given in a percentage from before anesthesia before and following anesthesia period over 60 min

SECONDARY OUTCOMES:
Proteome: overexpression of immune depressive proteins | 70-90 min
  Primary Outcome Measure:
  2.Overexpression of immune depressing proteins in the protein of maccrophages in in the 3-D- Gel electrophoresis as given in a percentage from before anesthesia before and following anesthesia period over 60 min

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Frietsch, Study Chair — University of Heidelberg, Faculty Mannheim